# Vale+Tú Salud: Corner-Based Randomized Trial to Test a Latino Day Laborer Program Adapted to Prevent COVID-19

NCT06146361

Version Date: 05/01/2023

#UTHealth Houston IRB NUMBER: HSC-SPH-20-1389 IRB APPROVAL DATE: 05/01/2023

### THE UNIVERSITY OF TEXAS HEALTH SCIENCE CENTER - HOUSTON

# VALE+Tú Salud: Corner-Based Randomized Trial to Test a Latino Day Laborer Program Adapted to Prevent COVID-19

## INFORMED CONSENT FOR VALE+ TÚ SALUD EXPERIMENTAL PARTICIPANTS

## **Dear Participant:**

The University of Texas School of Public Health is conducting "Vale+Tú Salud," a program to measure and address COVID-19 safety practices among Latino day laborers. We are inviting you to participate in a program to promote the implementation of COVID-19 safety practices that will include a 45-60-minute interview followed by a 30-45-minute group COVID-19 safety activity. Your total time commitment for this study won't exceed 2 hours. The purpose of the surveys is to learn about your beliefs and practices regarding the COVID-19 outbreak. The purpose of the safety activity is you assist you in developing a safety plan that you can easily implement to lower the COVID-19 risks for yourself and those around you. In addition, we are going to invite you to partner with us by sharing informational materials with the people in your social circles. All information materials will be provided by us free of charge in Spanish.

Four weeks after you complete the program, we will contact you by phone to conduct a follow up survey. By giving us your consent to participate in our study, you agree to participate in the initial survey, the COVID-19 safety activity, and the follow up assessment.

Your decision to take part in our study is voluntary, this means that you can refuse to answer any question you do not want to answer and there are no right or wrong answers to our questions. You may also stop your participation in the job safety activity at any point. Similarly, you can distribute as many flyers as you would like or not distribute any at all. The distribution of materials is optional and it won't affect your continued participation in the study. We also want to let you know that nobody will get upset if you do not answer a question, and nobody will deny you services as part of this program or at the University of Texas Health Science Center, if you refuse to participate in the survey or the activity.

A member of our research team will read aloud each question to you, and then record all of your answers on the iPad. We can pause the survey if you need to talk to a potential employer or are offered a job, and we will contact you at a later time if you want to finish the questions.

All of your answers will be stored in a secured computer and only study personnel with a password will be able to access them. All of your answers will be confidential. We will ask your name and contact information, and your contact information will only be collected, with your permission, in case you need to finish the survey or activity at a later time and to conduct the follow up survey. We will also request alternative contact information from people who might know your whereabouts in case we can't locate you. You can choose what contact information you would like to share with us. It is also okay if you don't want to share any contact information with us.

No one outside the study will have access to any information or comments you share with us today. This study has been granted a Certificate of Confidentiality by the National Institute of Health to give additional protection of your responses. The results of this survey will be presented as group information and your name will never be mentioned.

To our knowledge, there are no known risks that can result from your participation in this study besides someone accidentally disclosing confidential information, but our research team will take **ALL** the necessary measures to protect the information you share with us today. In addition, due to the current pandemic, additional safety measures are being taken to ensure your safety. All research staff will be wearing masks and other safety equipment. We will also provide you with a mask if you don't have one.

IRB NUMBER: HSC-SPH-20-1389 IRB APPROVAL DATE: 05/01/2023 Research staff and participants must observe social distance. Hand sanitizer will also be available to you for use throughout our COVID-19 safety activity.

Although, you will not benefit directly from participating in this survey, the information you share with us will help us refine the program to prevent the spread of COVID-19 that we will complete among Houston Latino day laborers. To compensate you for your time and valuable contributions to the Vale+Tú Salud program today, we will give you a gift card for \$50 after you complete the initial survey and the group activity. We will give you an additional \$75 gift card after completing the follow-up survey.

The Principal Investigator of this study is Dr. Maria Eugenia Fernandez-Esquer, who works at the School of Public Health at the University of Texas Health Science Center in Houston. If you want more information about this project, please call her at and she will gladly answer your questions.

You will receive a copy of this form to take home with you.

#### **CPHS STATEMENT**

This study (**HSC-SPH-20-1389**) has been reviewed by the Committee for the Protection of Human Subjects (CPHS) of The University of Texas Health Science Center at Houston. For any question regarding the investigation of the rights of the human subjects of the research, or to report an accident related to the research, call CPHS at \_\_\_\_\_\_\_.

I have read the information provided in this form, and I understand that my participation is completely voluntary.

By selecting the "Agree" button, I am agreeing to take part in this research study.

IRB NUMBER: HSC-SPH-20-1389
IRB APPROVAL DATE: 05/01/2023